CLINICAL TRIAL: NCT05706246
Title: Perioperative Hypersensitivity in Children; a Prospective Multidisciplinary Study
Brief Title: Perioperative Hypersensitivity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayca Kiykim, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HIPOP
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Drug Allergy
Keywords: children,; anesthesia; anaphylaxis
MeSH Terms: conditions — Drug Hypersensitivity; Anaphylaxis | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with perioperative hypersensitivity (Other): Children with perioperative hypersensitivity
  Interventions: Diagnostic Test: diagnostics

INTERVENTIONS:
Diagnostic Test: diagnostics — Serum tryptase levels were evaluated in all suspected children with perioperative hypersensitivity

SUMMARY:
There are limited studies on perioperative hypersensitivity (POH) reactions in children. The diagnosis of POH might be underestimated due to the difficulty of recognizing the reactions. Anaphylaxis may go unnoticed due to the unconscious state of the patient. Urticaria may be overlooked due to the sterile covers. This study aimed to evaluate POH reactions prospectively.

DETAILED DESCRIPTION:
Patients with intraoperative signs of diffuse erythema, urticaria, angioedema, sudden hypotension, tachycardia, bradycardia, arrhythmia, bronchospasm, vomiting, difficulty in ventilation, and end-tidal carbon dioxide (CO2) increase were included in the study. Reactions were graded from I to IV depending on increasing severity (Grade I, presence of cutaneous signs; Grade II, presence of measurable but non-life-threatening symptoms, including cutaneous effects, arterial hypotension, cough, or difficulty in mechanical ventilation; Grade III, presence of life-threatening reactions: cardiovascular arrest, tachycardia or bradycardia, arrhythmias, severe bronchospasm; Grade IV, circulatory inefficacy, cardiac and/or respiratory arrest).

In case of suspicious findings in terms of hypersensitivity reactions during surgery or recovery from anesthesia; the basal serum tryptase level was recorded at the time of the reaction, 2 hours after the reaction, and any time after 24 hours.

The severity of the reaction, vital signs, treatments applied, and medications administered after the reaction were recorded in the pre-prepared follow-up form. Then, skin tests were performed with all exposure agents,latex and chlorhexidine 4-6 weeks after the reaction in accordance with the records kept by the Pediatric Allergy and Immunology Clinic. A wheal diameter of at least 3mm larger than negative control is regarded a positive skin prick test, while in intradermal testing (IDT), a diameter 3 mm larger than the intracutaneously administered depot of the drug solution following 15-20 min is considered positive. Histamine was used as a positive control, and saline as a negative control. For positive skin test cases, basophil activation test was performed with the available drug. Skin prick and intradermal test concentrations were applied according to the recommendations for non-irritant test concentrations published by the European Network for Drug Allergy (ENDA) (8). Specific immunoglobulin E (spIgE) measurements were performed for latex and chlorhexidine on skin test positive cases, and for penicillin before the skin test for one case that experienced anaphylaxis due to antibiotics. The methodology used was ImmunoCAP® (Thermo Fisher Scientific, Uppsala, Sweden). Serum total tryptase levels were measured with ImmunoCAP® (Thermo Fisher Scientific). The increased serum tryptase value was calculated with the following formula: >1.2*basal tryptase level +2 mcg/L. In suspicious cases where the latex skin test was not clinically compatible, cutaneous provocation with latex was performed. Comparisons were made with the basophil activation test for positive results in drug skin tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intraoperative signs of diffuse erythema, urticaria, angioedema, sudden hypotension, tachycardia, bradycardia, arrhythmia, bronchospasm, vomiting, difficulty in ventilation, and end-tidal carbon dioxide (CO2) increase were included in the study.
* Children (0-18 years)

Exclusion Criteria:

* Refusing skin tests

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Perioperative hypersensitivity frequency | immediately after the reaction, within two hours following the reaction and basal tryptase levels

SECONDARY OUTCOMES:
Defining the culprit agent | 4 weeks after the reaction
  skin tests, specific immunoglobulin E levels and basophil activation tests were performed

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Kiykim, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No